CLINICAL TRIAL: NCT03195738
Title: Feasibility and Effects of the CO-OP Approach for Post-concussion Rehabilitation
Brief Title: Feasibility of a Cognitive Intervention for Youth Post Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Ontario Society of Occupational Therapists (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB14-485
Record Dates: First submitted 2017-06-14; First posted 2017-06-22 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Mild Traumatic Brain Injury; Concussion, Mild
Keywords: pediatrics; case series; feasibility
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): The Cognitive Orientation to Occupational Performance (CO-OP) Approach will be delivered over 10 30-60 minute sessions over a seven week period as follows: 2 sessions/week for 3 weeks, then 1 session per week for 4 weeks. In the CO-OP intervention participants are first assisted to identify 3-5 occupation based goals which will be the focus of the intervention sessions. Over the course of the 10 intervention sessions, participants are guided to learn and practice problem solving using a metacognitive strategy, "Goal-Plan-Do-Check" applied to their self-identified goals. Study therapists use 'guided discovery' an iterative technique to facilitate problem solving by the participant to develop plans to work toward their goals and to evaluate their progress. Intervention takes place in the location that is most meaningful for the participant's selected goal (e.g. home, school, playground etc.). Participants are provided with a work book to track progress.
  Interventions: Other: Cognitive Orientation to Occupational Performance (CO-OP)

INTERVENTIONS:
Other: Cognitive Orientation to Occupational Performance (CO-OP) — In the CO-OP intervention participants are first assisted to identify 3-5 occupation based goals which then become the focus of the intervention sessions. Over the course of the 10 intervention sessions, participants are guided to learn and practice problem solving using a metacognitive strategy, "Goal-Plan-Do-Check" applied to their self-identified goals. Study therapists use 'guided discovery' an iterative technique to facilitate problem solving by the participant to develop plans to work toward their goals and to evaluate their progress. Intervention takes place in the location that is most meaningful for the participant's selected goal (e.g. home, school, playground etc.). Participants are provided with a work book to track progress.

SUMMARY:
The purpose of this study is to evaluate the feasibility and effects of a cognitive intervention for youth following concussion

DETAILED DESCRIPTION:
Concussion, a form of mild traumatic brain injury, is one of the most commonly reported injuries in youth. While most recover quickly, a substantial subset (30-58.5%) report symptoms that persist at one month with a reported 11-14% who continue to report symptoms beyond three months. Currently, there are no evidence-based guidelines for treatment that address occupational (meaningful activity) concerns for youth who are slower to recover post-concussion. It is postulated that a top-down rehabilitation approach with metacognitive strategy training as the core of the intervention might be effective.The Cognitive Orientation to Occupational Performance (CO-OP) Approach is a metacognitive strategy training approach with a growing body of literature supporting it's value in improving participation in meaningful activity and achieving self-selected occupation-based goals for adults with brain injury and youth with moderate to severe brain injury.Given the long-term occupational concerns in youth with persistent post-concussion symptoms, and the lack of evidence based interventions for these youth, it is hypothesized that the CO-OP Approach may facilitate return to meaningful occupation in this population.

ELIGIBILITY:
Inclusion Criteria:

* concussion diagnosed by a physician;
* presence of at least one post-concussion symptom for three months or more; -experiencing challenges with usual daily activities secondary to post-concussive symptoms;
* able to identify four or more occupation-based goals;
* 12-18 years of age;
* no concurrent serious medical or psychiatric diagnoses.
* has a parent who can support participation and participate in a post intervention interview

Exclusion Criteria:

* non English speaking

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2014-07-25 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Occupational Performance and Satisfaction (Canadian Occupational Performance Measure) | Measure will be administered at baseline, within one week post intervention (i.e. at 8 weeks) and again at 3 month follow up.
  A change score of two points is considered clinically significant (McColl, Carswell, Law, Pollock, Baptiste, & Polatajko 2006). During a semi-structured interview, clients are asked to identify a minimum of five occupational performance issues (OPI's). The five most important OPI's as determined by the client are identified using a ranking scale (1=not important at all to 10=extremely important) and then ranked according to performance and satisfaction with performance using 10 point scales (Performance score of 1=not able to do it to 10=able to do it extremely well; Satisfaction score of 1=not at all satisfied to 10=extremely satisfied).

SECONDARY OUTCOMES:
Change in mood and self-concept (Beck Youth Inventories) | Measure will be administered at baseline, within one week post intervention (i.e. at 8 weeks) and again at 3 month follow up.
  The Beck Youth Inventories for children and adolescents-Second Edition (BYI-II) (Beck, Beck, Jolly, & Steer, 2005) provides insight into youth's negative thoughts about their self, life and future, and feelings of sadness, worry, guilt, anger, disruptive behaviors and self-worth. The depression, anxiety and anger inventories were administered. Higher scores are associated with negative affect. Psychometric properties are strong with high internal consistency (Cronbach's alpha coefficients from .91-.96) and test-retest reliability (r=.83 to .93).
Change in symptoms (Post Concussion Symptom Inventory) | Measure will be administered at baseline, within one week post intervention (i.e. at 8 weeks) and again at 3 month follow up.
  The 22-item Post-Concussion Symptom Inventory (PCSI) (Sady, Vaughan, Gioia, 2014) (adolescent version) measures the presence and severity (on a scale of 1 (not a problem)-6 (severe problem)) of concussion symptoms. The PCSI has moderate to good inter-rater reliability (r=0.4 to r=0.5), test-retest reliability (r=0.62 to 0.84) and internal consistency (r=0.72 to 0.93). Higher scores indicate presence of more/worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Anne W Hunt, PhD, Principal Investigator — Bloorview Research Institute
Locations (1):
- Bloorview Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Law, M., Baptiste, S., Carswell, A., McColl, M., Polatajko, H., & Pollack N. (2014). Canadian Occupational Performance Measure (5th ed.). Ottawa: CAOT Publications.
- [Background] McColl, MA., Carswell, A., Law, M., Pollock, N., Baptiste, S., & Polatajko, H. (2006). Research on the Canadian Occupational Performance Measure: an annotated resource. Ottawa: CAOT Publications.
- [Background] Sady MD, Vaughan CG, Gioia GA. Psychometric characteristics of the postconcussion symptom inventory in children and adolescents. Arch Clin Neuropsychol. 2014 Jun;29(4):348-63. doi: 10.1093/arclin/acu014. Epub 2014 Apr 15. PMID 24739735
- [Background] Beck, J., Beck, A., Jolly, J., & Steer, R. (2005). Beck Youth Inventories for Children and Adolescents. 2nd Ed. San Antonio: Harcourt Assessment Inc.